CLINICAL TRIAL: NCT07140887
Title: Autogenous Bone Ring Versus Split Bone Block With Simultaneous Implant Placement for Management of Posterior Atrophic Mandible (A Randomized Clinical Trial)
Brief Title: Autogenous Bone Ring Versus Split Bone Block for Management of Posterior Atrophic Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0917-05/2024
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Ridge Augmentation
Keywords: Bone ring, trephine, piezotome, ridge augmentation, Khoury technique, implant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone ring technique (Experimental)
  Interventions: Other: Bone Ring
- Split bone block technique (Active Comparator)
  Interventions: Other: Split Bone block

INTERVENTIONS:
Other: Bone Ring — Patients in this group will be treated with the bone ring technique. An implant drill will be used next to prepare central osteotomies corresponding to the final implant diameter to be placed in the center of the disc converting it to a "bone ring".
  Arms: Bone ring technique
Other: Split Bone block — Patients of this group will be treated with split bone block with simultaneous implant technique. The bone shell will be split into two bone shells each 1 ~ 2 mm in thickness using a disc.
  Arms: Split bone block technique

SUMMARY:
Teeth loss in the posterior mandible initiates residual ridge resorption especially in vertical direction, this causes difficulty in implant placement so ridge augmentation must be done either simultaneous with implant placement or in a staged approach Aim: To evaluate the effect of bone ring technique versus split bone block technique with simultaneous implant clinically on primary and secondary

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing posterior mandibular teeth.
* Vertical bone defect from 3 to 4 mm.
* Adequate zone of keratinized tissue.

Exclusion Criteria:

* Presence of infection or periapical lesions in adjacent teeth.
* Medically compromised patients with a condition that affects the procedure.
* Insufficient inter-arch distance.
* Bruxism or clenching.
* Alcoholism.
* Heavy Smokers.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | Immediate and 6 months
  Implant stability will be recorded immediately after placement (1ry stability) and after 6 months (2ry stability ) by using osstell device. The result is presented in form of ISQ value from 1to 100, the higher the ISQ the higher the stability of implant(
Change in pain scores | up to 7 days
  Pain will be assessed for 7 days postoperatively using 10-point visual analouge scale (VAS) (0-1=None, 2-4=mild, 5-7=moderate, 8-10=severe ).
Change in marginal bone level | 6 and 9 months
  At buccal, lingual, mesial, and distal sites will be evaluated radiographically from the shoulder of the implant to the alveolar crest.

SECONDARY OUTCOMES:
Change in bone density | 6 months
  Will be measured at 6 points around the implant and a mean value will be calculated using CBCT
Change in edema | up to 7 days
  Measured as follows:
  No inflammation = none. Intra oral swelling confined to the surgical field = mild. Extra oral swelling in the surgical zone =moderate. Extra oral swelling spreading beyond the surgical zone =intense.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt